CLINICAL TRIAL: NCT06751225
Title: Evaluation of Wear Experience With a Weekly Replacement Soft Contact Lens in Neophyte Lens Wearers With Astigmatism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Jennifer Fogt, Assistant Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024H0379
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Astigmatism Bilateral

STUDY DESIGN:
Intervention Model Description: Subjects will be fit into the one week replacement soft contact lens to wear for 3 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Contact Lens Wear Experience (Experimental): One week replacement soft contact lenses will be worn for 3 weeks.
  Interventions: Device: One week replacement soft contact lenses

INTERVENTIONS:
Device: One week replacement soft contact lenses — One week replacement soft contact lenses

SUMMARY:
This open-label study is of adults with astigmatism who have never worn contact lenses. Subjects will be fit into a one week planned-replacement contact lenses and will wear lenses for approximately 3 weeks. Subjects will return for vision and lens fit assessments and will complete surveys about their wear experience.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be new to contact lenses and have astigmatism of -0.75 or greater (within the parameters available for the P7fA lenses)
2. Subjects must have 20/20 or better best corrected visual acuity.
3. Good general health (defined by medication use that has not changed within the last month and the absence of medical conditions or treatments that are deemed confounding to the data as determined by the PI)
4. Ability to give informed consent
5. Willing to spend time for the study. Subjects will be required to attend three study visits and wear contact lenses on days between study visits.
6. Willing and able to wear contact lenses for at least 8 hours per day for 5 days per week during the study as daily wear.
7. Currently not using eye lubricating drops and willing to not use during study.
8. Either gender and 18-40 years of age.
9. Any racial or ethnic origin

Exclusion Criteria:

1. Any active ocular inflammation or infection.
2. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable.
3. Are presbyopic and require or habitually uses reading glasses for near work
4. Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable
5. History of refractive surgery
6. Meets the diagnosis of dry eye disease with OSDI screening score ≥13.
7. Known history of allergy or sensitivity to contact lens solutions and/or sodium fluorescein
8. Is pregnant or lactating or planning a pregnancy during enrollment in the study
9. Is participating in another clinical research study that includes invasive ocular tests
10. An inability to perform contact lens application and removal after instruction.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Subjective assessment of lens wear experience | 3 weeks
  VAS assessment of overall vision throughout the day. (0-100 scale; 0=unacceptable 100=excellent)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University College of Optometry, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No